CLINICAL TRIAL: NCT01209390
Title: A Prospective, Open Label, Multi-centre, Post-marketing Registry on the Use of ChondroMimetic for the Repair of Osteochondral Defects
Brief Title: A Prospective, Post-marketing Registry on the Use of ChondroMimetic for the Repair of Osteochondral Defects
Acronym: OMCM
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment rate
Sponsor: TiGenix n.v. (Industry)
Responsible Party: Sponsor
Other Study IDs: OMCM-2010-01
Record Dates: First submitted 2010-08-06; First posted 2010-09-27 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Osteochondral Defects
Keywords: osteochondral; regenerative; repair; cartilage lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteochondral lesions: Patients with osteochondral lesions in the knee, the ankle, or other joint
  Interventions: Device: Chondromimetic

INTERVENTIONS:
Device: Chondromimetic — The Chondromimetic implant is intended to serve as a scaffold for cellular and tissue ingrowth in osteochrondral defect repair such as bone and/or cartilage.
  The plug consists of a chondral layer with collagen and GAG and an osseus layer with collagen, GAG, and calcium phosphate.
  Other Names: Osteochondral repair plug; CM

SUMMARY:
The objective of this post-marketing study is to confirm the clinical efficacy and safety outcome of treatment with ChondroMimetic in a patient population within the proposed indication (osteochondral cartilage defects), over a 36 months post-implantation follow-up period.

The primary objective is to collect post-marketing safety data in a real life setting by means of (S)ADR reporting.

The secondary objectives are:

* Clinical outcome as assessed by patient reported EuroQoL-5D
* Structural repair as assessed by MRI
* The number of treatment failures and the time to treatment failure
* The ease of use of ChondroMimetic as reported by the surgeon

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient informed consent
2. Shallow osteochondral defect ≤ 12 mm diameter and ≤ 8 mm depth in weight bearing area
3. Agree to actively participate in a rehabilitation protocol

Exclusion Criteria:

1. Severe vascular or neurological disease
2. Uncontrolled diabetes
3. Severe degenerative joint disease
4. Pregnancy
5. Presence of infection at the site or in the joint space (e.g. osteomyelitis)
6. Diagnosis rheumatoidism
7. Advanced osteoarthritis as judged by the surgeon
8. Drug and/or alcohol abuse
9. Hypercalcemia
10. Known allergy to any of the components of the device (e.g. bovine collagen)
11. Bleeding disorders of any etiology
12. Steroidal or immunosuppressive maintenance therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in selected centres, primary or secondary care, first line or referral treatment.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Safety data | on ongoing basis up to 3 years
  Safety data as measured by adverse device reactions

SECONDARY OUTCOMES:
EuroQoL-5D | baseline, 6, 12, 24, 36 months
  The EQ-5D is a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension
MRI | baseline, 12, 24, 36 months
  Structural repair will be assessed by MRI. The available MRIs will be collected and scored by an independent radiologist, using the published MOCART score , and one additional item, level of the subchondral bone plate.
Failure rate | 3 years
  Treatment failure is defined as "a re-intervention on the index lesion, prompted by persistence or recurrence of symptoms related to the index knee". The date of failure is the actual date of re-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Hangody, MD, Principal Investigator — Uzsoki Hospital, Budapest, Hungary
Locations (4):
- University Hospitals Leuven, Leuven, Belgium
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany
- Uzsoki Hospital, Budapest, Hungary
- Addenbrookes Hospital, Cambridge, United Kingdom